CLINICAL TRIAL: NCT00527852
Title: Assessment of Flocked Swabs for the Identification of Group A Streptococcal Pharyngitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: David Goldfarb, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 07/59X
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2007-07

CONDITIONS: Streptococcal Infection; Pharyngitis
Keywords: Flocked swab; Group A streptococcus pharyngitis
MeSH Terms: conditions — Streptococcal Infections; Pharyngitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Flocked swab

SUMMARY:
This is a study to to compare traditional fibre wound swabs to more recently developed flocked swabs for the identification of Group A streptococcal pharyngitis in children presenting to a children's emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Need for a bacterial throat culture

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Identification of Group A streptococcus via culture of organism

CONTACTS AND LOCATIONS:
Overall Officials: David M Goldfarb, MD FRCPC, Principal Investigator — Children's Hospital of Eastern Ontario, Division of Infectious Disease
Locations (1):
- Children's Hospital of Eastern Ontario Emergency Department, Ottawa, Ontario, Canada